CLINICAL TRIAL: NCT05078619
Title: Percutaneous Coronary Intervention Before Transcatheter Aortic Valve Implantation: the PRO-TAVI Trial
Brief Title: Percutaneous Coronary Intervention Before Transcatheter Aortic Valve Implantation
Acronym: PRO-TAVI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Michiel Voskuil, MD, PhD, Professor in Cardiology, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL77915.041.21
Record Dates: First submitted 2021-09-21; First posted 2021-10-14 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Valvular Heart Disease; Aortic Valve Stenosis; Coronary Artery Disease
Keywords: Transcatheter aortic valve implantation; Percutaneous coronary intervention
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAVI without routine PCI (Experimental): Patients who are randomized to the experimental or index group undergo TAVI without routine PCI
  Interventions: Procedure: No PCI
- TAVI with routine PCI (No Intervention): Patients who are randomized to the control or reference group undergo TAVI with routine PCI

INTERVENTIONS:
Procedure: No PCI — Omission of PCI of significant coronary artery disease prior to TAVI
  Arms: TAVI without routine PCI

SUMMARY:
The aim of this trial is to evaluate the safety and cost effectiveness of omission of percutaneous coronary intervention of significant coronary artery disease in patients scheduled to undergo transcatheter aortic valve implantation.

ELIGIBILITY:
Inclusion Criteria:

* Severe AoS meeting the criteria stated by the ESC in the ESC/EACTS Guidelines for the management of valvular heart disease AND considered symptomatic (NYHA functional class ≥ 2);
* TAVI decided by multidisciplinary Heart Team taken into account the international standards by ESC and guidelines of Dutch Society for Cardiology (NVVC);
* ≥ 1 stenosis in epicardial coronary artery (> 2.5mm) or bypass graft. Stenosis is considered significant if angiographic 70-99% or angiographic 40-70% with positive hemodynamic parameters.
* Written informed consent.

Exclusion Criteria:

* Unprotected LM-stenosis or equivalent
* No PCI-eligible stenosis
* Contraindication for DAPT
* Life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
composite of all-cause mortality, myocardial infarction, stroke and type 2-4 bleeding, in accordance to VARC-3 criteria | 12 months from randomization

SECONDARY OUTCOMES:
Composite of all-cause mortality, myocardial infarction, stroke, in accordance with VARC-3 criteria | 4 months - 12 months - total follow up 5 years
all-cause mortality | 4 months - 12 months - total follow up 5 years
  VARC-3
myocardial infarction | 4 months - 12 months - total follow up 5 years
  VARC-3
stroke | 4 months - 12 months - total follow up 5 years
  VARC-3
VARC-3 bleeding | 4 months - 12 months - total follow up 5 years
BARC bleeding | 4 months - 12 months - total follow up 5 years
  BARC bleeding > type 1
urgent and elective revascularization | 4 months - 12 months - total follow up 5 years
  ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials & ARC-2
Target lesion revascularization | 4 months - 12 months - total follow up 5 years
  ARC-2
Target vessel revascularization | 4 months - 12 months - total follow up 5 years
  ARC-2
rehospitalization | 4 months - 12 months - total follow up 5 years
  VARC-3
Left ventricular function measured by echocardiography | 12 months
Cost-effectiveness of omission of PCI using QALYs | 4 months - 12 months
Cost-effectiveness of omission of PCI using Incremental Cost Effectiveness Ratios | 4 months - 12 months
Quality of life assessed by Euro Quality of Life 5D Questionnaire | 4 months - 12 months
  the system produces a 5-digit health status profile to describe quality of life in a descriptive manner. Therefore, no lowest and highest value can be stated.
Quality of life assessed by SF-36 Questionnaire | 4 months - 12 months
  Questionnaire consists of eight sections. Each section is transformed into a 0 - 100 scale. The lower the score the more disability.
Anginal status (CCS) | 4 months - 12 months
NYHA classification | 4 months - 12 months
Acute kidney injury stage 3 and 4 | 4 months - 12 months - total follow up 5 years
  VARC-3

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Voskuil, MD PhD, Principal Investigator — UMC Utrecht
Locations (12):
- Netherlands (12):
  - RadboudUMC, Nijmegen, Gelderland
  - Maastricht UMC+, Maastricht, Limburg
  - Amphia Ziekenhuis Breda, Breda, North Brabant
  - Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland
  - OLVG, Amsterdam, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - UMC Groningen, Groningen, Provincie Groningen
  - Haga Ziekenhuis Den Haag, The Hague, South Holland
  - Antonius Ziekenhuis Nieuwegein, Nieuwegein, Utrecht
  - UMC Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aarts HM, Hemelrijk KI, Broeze GM, van Ginkel DJ, Versteeg GAA, Overduin DC, Tijssen JG, Beijk MAM, Baan J, Vis MM, Lemkes JS, de Winter RJ, Dickinson MG, Kraaijeveld AO, Mokhles MM, Dessing TC, Grundeken MJ, Claessen BEPM, Tonino PAL, Schotborgh CE, Meuwissen M, van Houwelingen GK, Wykrzykowska JJ, Amoroso G, Vossenberg TN, Vriesendorp PA, van Royen N, Ten Berg JM, Delewi R, Voskuil M. Deferral of routine percutaneous coronary intervention in patients undergoing transcatheter aortic valve implantation: Rationale and design of the PRO-TAVI trial. Am Heart J. 2025 Mar;281:133-139. doi: 10.1016/j.ahj.2024.12.003. Epub 2024 Dec 16. PMID 39674524